CLINICAL TRIAL: NCT02263365
Title: Prospective Randomized Control Study on Effect of Post Operative Loperamide in Decreasing Readmission for Dehydration in Colorectal Patients After Diverting Ileostomies
Brief Title: Use of Post Operative Loperamide in Colorectal Patients After Diverting Ileostomies
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to meet study requirements
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Phillip Fleshner MD, Director of Colorectal Residency, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Loperamide Dehydration
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Results first posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-11

CONDITIONS: Dehydration, Diverting Ileostomy, Loperamide
MeSH Terms: conditions — Dehydration | interventions — Loperamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Therapeutic (Experimental): Patients randomized to this arm will be administered 4mg tid (three times daily) of loperamide from the day of discharge onwards. A total of duration of 14 days of medication will be administered
  Interventions: Drug: Loperamide

INTERVENTIONS:
Drug: Loperamide — Loperamide 12mg per day (4mg t.i.d) for 2 weeks post discharge
  Arms: Therapeutic

SUMMARY:
Dehydration post creation of a diverting ileostomy is a common and debilitating problem faced by patients undergoing ileal-anal pouch anastomoses for both inflammatory bowel disease and familial adenomatous polyposis (FAP) syndrome. Those patients with low rectal cancers or other polyposis syndromes e.g. HNPCC hereditary non polyposis colorectal cancers, may potentially have a delay in the adjuvant therapy when faced with this complication.

Studies performed in this groups of patients report a readmission rate of 17-21% for dehydration.

Loperamide has been shown to significantly decrease the daily volume of weight of stool in these patients.

The purpose of this study is to establish whether loperamide given at 4mg three times daily for 14 days from day of discharge empirically decreases 30 days readmission rate for dehydration.

The investigators hypothesize that there will be a 15% decrease from 25% to 10% in the readmission rates, that severity of dehydration will be decreased.

ELIGIBILITY:
Inclusion Criteria:

1. Able to freely give written informed consent to participate in the study and have signed the Informed Consent Form;
2. Males or females, age 18 and older at the time of study screening;
3. American Society of Anesthesiologists (ASA) Class I-III (Appendix III) undergoing elective surgery

Exclusion Criteria:

1. Mentally incompetent or unable or unwilling to provide informed consent or comply with study procedures
2. American Society of Anesthesiologists (ASA) Class IV or V; emergency surgeries
3. Children <18
4. Pregnant patients
5. Patients who have intra-abdominal sepsis or partial or intermittent bowel obstruction or enteritis
6. Patients who are on long term steroids, opioids or antidiarrheals pre operatively
7. Patients who are administered pro kinetics eg. Metoclopramide
8. Patients with recurrent disease in their small bowel - Crohn's disease, or previous irradiated pelvis resulting in irradiation bowel disease
9. End ileostomies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10-07 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip R Fleshner, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: No intervention
Period: Overall Study
Arm/Group | Control | Therapeutic
Started | 22 | 18
Completed | 0 | 0
Not Completed | 22 | 18
Not completed — Physician Decision | 22 | 18

BASELINE CHARACTERISTICS:
Population: Data was not collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Therapeutic | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of 30 Day Readmission (Severe Dehydration)
Time Frame: 30 day
Population: Data was not collected.
Arm/Group | Control | Therapeutic
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Moderate Dehydration Resulting in Outpatient Visits or ER Intervention That is =/<24hrs That Did Not Require Hospital Admission
Time Frame: 30 day
Population: Data was not collected.
Arm/Group | Control | Therapeutic
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Mild Dehydration - Subjective Report of Difficulty in Managing Fluid Balances and Stoma Care
Time Frame: 30 days
Population: Data was not collected.
Arm/Group | Control | Therapeutic
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Length of Index Admission
Time Frame: 30 day
Population: Data was not collected.
Arm/Group | Control | Therapeutic
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Data was not collected. Study was terminated prematurely due to issued with compliance. Total number of participants at Risk (e.g., " All-Cause Mortality, Serious, and other [not including serious] adverse events were not monitored/assessed for this study.
Arm/Group | Control | Therapeutic
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study only accrued 40 patients. Due to issues with enrollment and study procedures compliance it was decided to terminate the study. Data analysis will not be done for this study. This study has been closed with the internal review board.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No